CLINICAL TRIAL: NCT00709410
Title: Mass Oral Cholera Vaccination in High-risk Populations in Zanzibar: Assessment of Effectiveness and Herd Protection
Brief Title: Mass Oral Cholera Vaccination in Zanzibar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Vaccine Institute (Other)
Collaborators: Ministry of Health and Social Welfare, Zanzibar (Other Government); National Institute of Cholera and Enteric Diseases, India (Other); Bill and Melinda Gates Foundation (Other); World Health Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DK - 02
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Cholera; Diarrhea
Keywords: Cholera, Diarrhea, Vaccination, Vaccines
MeSH Terms: conditions — Cholera; Diarrhea | interventions — Dukoral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): This is a single arm study. All consenting, eligible participants will receive the oral cholera vaccine.
  Interventions: Biological: rBS-WC vaccine

INTERVENTIONS:
Biological: rBS-WC vaccine — 1 mg of recombinant cholera toxin B subunit and approximately 1 x 10^11 of inactivated whole cells of Vibrio cholerae O1 Inaba and Ogawa, classic and El Tor strains (6). The rBS-WC vaccine is supplied as 3 ml single-dose vials each with a sachet of sodium bicarbonate buffer. Buffer solution will be prepared by dissolving the sachets in drinking water (150 ml water for each sachet of sodium bicarbonate). The full dose of vaccine will be mixed with 40, 75, or 150 ml of buffer solution for persons 2 to 4 years, 5 to 11 years, and over 11 years old, respectively. The vaccine is recommended to be given in two doses with an interval of at least seven days and protection is conferred 7 to 10 days after the second dose.
  Other Names: Dukoral™

SUMMARY:
The purpose of this study is to conduct cholera vaccinations in high-risk populations in Zanzibar in order to estimate herd protection conferred by the vaccine,estimate effectiveness of the vaccine, and describe the interaction of vaccination and improved water supply on the burden of cholera and diarrhoeal diseases.

DETAILED DESCRIPTION:
The seventh cholera pandemic began in Indonesia in 1961 and spread quickly to other Asian countries. In 1970, the etiologic agent, Vibrio cholerae O1 El Tor, invaded sub-Saharan Africa, whose residents had not experienced cholera for more than 100 years. Outbreaks rapidly occurred and the disease has become endemic in several parts of the continent. In 2006, Africa reported 234,349 cholera cases to the WHO, accounting for 99% of the officially-notified global cholera (1). Between 1995 and 2005, 66% of cholera outbreak reports to ProMed came from sub-Saharan Africa (2). There is growing evidence of the large and increasing burden of cholera in Africa.

One African country that is severely and repeatedly affected by cholera is Zanzibar. After the first case of cholera was confirmed in the country in January 1978, regular outbreaks have been reported (3). These outbreaks cause human suffering, are socially disruptive, and divert resources from other essential services. Cholera control in Zanzibar has focused mainly on case management, water chlorination campaigns, and dissemination of hygiene messages. The Ministry of Health and Social Welfare (MOHSW) is eager to identify new and effective tools, such as oral cholera vaccination, that could be implemented in Zanzibar.

In 2002, the World Health Organization (WHO) recommended the potential use of oral cholera vaccines in endemic and epidemic situations, but it was deemed necessary to gain more experience through demonstration projects (4). Since then, mass oral cholera vaccinations have been conducted in Beira, Mozambique (5), in Darfour, Sudan, and in Aceh, Indonesia which demonstrated the feasibility and effectiveness of vaccination under actual public health conditions. The only oral cholera vaccine available in the market consists of killed whole-cell V. cholerae O1 with purified recombinant B-subunit of cholera toxin (WC/rBS) administered with a buffer solution as two doses, at least a week apart. The vaccine is internationally-licensed (including in Zanzibar) for use in individuals 2 years of age and older. This vaccine, and its predecessor (BS-WC) that contained chemically extracted rather than recombinant cholera toxin B subunit, have been shown to be safe and protective in several trials conducted in cholera-endemic settings in Asia and South America (6-9) and in a sub-Saharan African setting with a high prevalence of HIV (5).

An incompletely answered question regarding this vaccine is its potential to confer herd protection (10). The level of herd immunity would determine the minimum vaccine coverage required to produce widespread protection against cholera in a community. A recent study comparing cholera rates in sites in Asia and Africa has shown that the burden of cholera is greatest in young children (11); herd immunity would provide protection for children too young to receive the vaccine, as well as other unvaccinated members of the community. Although recent re-analysis of data from the large placebo-controlled field trials of the oral cholera vaccine in Bangladesh in the 1980s showed substantial herd protection from vaccination (12,13), there may be limitations to the applicability of these findings to other cholera endemic settings with different living conditions (14). Mathematical modelling of the same Bangladesh data found that cholera transmission could be controlled in endemic areas with 50% vaccine coverage. At this level of coverage, the model predicted that there would be an 89% reduction in cholera cases among the unvaccinated, and a 93% reduction overall in the entire population. A more modest coverage of 30% would result in a 76% reduction in cholera incidence for the population area covered (15). If confirmed in actual field studies, these mathematical predictions have major vaccine cost-effectiveness implications.

We propose to carry out mass oral cholera vaccinations in populations at high risk for cholera in Zanzibar followed by an assessment of direct and indirect protection. The WHO was awarded a grant by the Bill and Melinda Gates Foundation entitled: "Pre-emptive use of a cholera vaccine in vulnerable populations at risk", under which this proposal will be funded. The 6 million US$ grant aims to address issues regarding the potential utilization and mechanism of pre-emptive delivery of the vaccine to prevent outbreaks in endemic regions. An important component is the potential creation of a "revolving" stock of vaccine and the financial sustainability of maintaining such a stockpile.

The lessons learned from this project will be crucial for informed decisions about the potential wider use of cholera vaccination in Zanzibar and other cholera-endemic sub-Saharan African countries. The lessons learned from the effectiveness study will form part of the evidence for the possible establishment of a sustainable vaccine stockpile. The project would provide essential information on the vaccine coverage required to control cholera in endemic areas and additional data on vaccine effectiveness in a different setting in Africa.

ELIGIBILITY:
Inclusion Criteria:

* Healthy residents of selected vaccination sites
* Aged 2 years and older
* non-pregnant

Exclusion Criteria:

* Age less than 2 years
* Pregnant

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 51151 (Actual)
Dates: Start 2009-01; Primary Completion 2009-02 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Receipt of 2 complete or nearly complete swallowed doses of oral cholera vaccine | after completion of the vaccination campaign

SECONDARY OUTCOMES:
Acute, non-bloody diarrhoea severe enough to seek care at the Primary Health Care Units | starting 10 days following vaccination campaign

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Khatib, MD, Principal Investigator — Ministry of Health and Social Welfare, Zanzibar
Locations (1):
- Ministry of Health and Social Welfare, Zanzibar, Zanzibar, Tanzania

REFERENCES:
- [Derived] Khatib AM, Ali M, von Seidlein L, Kim DR, Hashim R, Reyburn R, Ley B, Thriemer K, Enwere G, Hutubessy R, Aguado MT, Kieny MP, Lopez AL, Wierzba TF, Ali SM, Saleh AA, Mukhopadhyay AK, Clemens J, Jiddawi MS, Deen J. Effectiveness of an oral cholera vaccine in Zanzibar: findings from a mass vaccination campaign and observational cohort study. Lancet Infect Dis. 2012 Nov;12(11):837-44. doi: 10.1016/S1473-3099(12)70196-2. Epub 2012 Sep 4. PMID 22954655
- [Derived] Hashim R, Khatib AM, Enwere G, Park JK, Reyburn R, Ali M, Chang NY, Kim DR, Ley B, Thriemer K, Lopez AL, Clemens JD, Deen JL, Shin S, Schaetti C, Hutubessy R, Aguado MT, Kieny MP, Sack D, Obaro S, Shaame AJ, Ali SM, Saleh AA, von Seidlein L, Jiddawi MS. Safety of the recombinant cholera toxin B subunit, killed whole-cell (rBS-WC) oral cholera vaccine in pregnancy. PLoS Negl Trop Dis. 2012;6(7):e1743. doi: 10.1371/journal.pntd.0001743. Epub 2012 Jul 24. PMID 22848772